CLINICAL TRIAL: NCT04726293
Title: Anti-inflammatory Effect and Associated Mechanisms of Mango Consumption in At-risk Overweight and Obese Population With Chronic Low-grade Inflammation
Brief Title: Anti-inflammatory Effect and Associated Mechanisms of Mango Consumption
Acronym: MG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-2020-57
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Overweight or Obesity; Healthy
Keywords: mango; Inflammatory markers; Gut microbiome; Metabolic responses
MeSH Terms: conditions — Overweight; Obesity | interventions — Mangifera indica extract

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango beverage (Experimental): Mango composite served as a frozen drink
  Interventions: Dietary Supplement: Mango
- Control beverage (Placebo Comparator): Energy matched Control frozen drink
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Mango — Mango beverage -1 cup fresh mango equivalent, twice a day for 4 weeks
  Arms: Mango beverage
Dietary Supplement: Control — control beverage 1 cup, twice a day for 4 weeks
  Arms: Control beverage

SUMMARY:
The primary objective of this project is to provide new knowledge through a comprehensive set of analyses that investigate the complex interplay between regular mango intake, gut microbial structure/ function, mechanisms of inflammation and insulin sensitivity in over weight (OW)/obese (OB) human subjects with chronic low-grade inflammation.

DETAILED DESCRIPTION:
The proposed study is a randomized, 2-arm, parallel, placebo-controlled design Human participants (n=44) with BMI >25 and high sensitivity C-Reactive Protein (hs-CRP), a global marker of inflammation, >1.0 and ≤10 ng/L will be recruited. Recruited subjects must meet all eligibility criteria, sign and date a written Institutional Review Board (IRB)-approved Informed Consent Form. Participants will be randomized into one of the two beverage intervention groups i.e., mango or control beverage.

Each subject will be asked to come for 1 Screening Visit, 1 pre-study, and 3 Test Day Visits (two of which will also include OGTT testing). The initial screening visit will provide subjects with their site-specific, IRB-approved informed consent document prior to the start of any study-related procedures. Subject eligibility will be determined through a high sensitivity C-Reactive Protein (hs-CRP) marker value, anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey related to general eating, health, mood and exercise habits.

Eligible subjects will follow a limited polyphenolic diet throughout the duration of their participation, although stricter guidelines will be imposed during the 3 days prior to a study visit that involved blood/urine/fecal collection. Shopping lists and meal plans will be provided to subjects, along with counseling by the study investigators, to help subjects adhere to the limited polyphenolic diet. The trial will initiate with a 3-day food diary to assess background (pre-study) dietary intake followed by counseling to follow a diet relatively low in (poly)phenolic rich-beverages/foods, which will be maintained for the duration of the experiment. After an initial 7-day wash-in period on the limited polyphenolic diet, subjects will be randomized to 1 of 2 test treatments based on a randomization schedule.

The three main Test Day visits will occur at Day 0; baseline), Day 14 (mid-point), and Day 28 (end-point). Two of the Test Day Visits(Day0 and Day 28) will last about 2.5-3 h and involve blood pressure (BP) measurements, anthropometric (weight, waist circumference; body composition) assessment, and an oral glucose tolerance test (OGTT) will be performed. The Test Day Visit on Day 14 will last about 1-1.5 hours, and subjects will be required to remain at the Clinical Nutrition Research Center for the duration of the visit. Fasting blood samples will be collected via a butterfly needle placed by a certified phlebotomist. Subjects will maintain daily food and GI-tract diary during the 4-week feeding trial. The diary will include questions about food intake and the condition of gastrointestinal tolerance and bowel function. Urine and fecal samples will be collected to monitor modifications occurring in the metabolites during the supplementation. .

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 20-60 years of age, inclusive with high sensitivity C-Reactive Protein (hs-CRP), a global marker of inflammation, >1.0 and ≤10 ng/
* BMI ≥ 25 kg/m2
* Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 2 years
* Judged to be in good health on the basis of the medical history ie., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food diary and GI tract questionnaire, sample collection and study visit schedule)
* Able to maintain usual physical activity pattern
* Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during study visit

Exclusion Criteria:

* Men and women who smoke
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at screening visit
* Men and women who have fasting blood glucose concentration >125 mg/dL at screening visit
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Men and women who are taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti inflammation, lipid lowering medication, blood pressure lowering medication, etc... - - Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
* Men and women who have participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator.
* Men and women who have used antibiotics within the previous 2 months
* Men and women who had gastrointestinal barium opaque meal within 3 months
* Men and women who used prebiotics, probiotics, or drugs active on gastrointestinal motility, or a laxative of any class within 1 month
* Men and women with history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Men and women who had substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d)
* Men and women who have donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Men and women who have unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Men and women who have unusual working hours i.e., working overnight (e.g. 3rd shift)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Characterize indices of systemic inflammation (IL-6) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim will include analysis of systemic markers of inflammation (IL-6) in plasma
Characterize indices of systemic inflammation mechanism of action after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim via Toll like receptor, Nuclear factor erythroid 2-related factor 2, and nuclear factor kappa-light-chain-enhancer of activated B cells (TLR/Nrf2/NF-κB) activation in Monocytes isolated from peripheral blood.
Characterize indices of systemic inflammation mechanism of action (Toll like receptor) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim via Toll-like receptor, activation in Monocytes isolated from peripheral blood.
Characterize indices of systemic inflammation mechanism of action (nuclear factor kappa-light-chain-enhancer of activated B cells ) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim via nuclear factor kappa-light-chain-enhancer of activated B cells activation in Monocytes isolated from peripheral blood.
Characterize indices of systemic inflammation mechanism of action (Nuclear factor erythroid 2-related factor 2) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim via (Nuclear factor erythroid 2-related factor 2 activation in Monocytes isolated from peripheral blood.
Characterize the gut microbiota in response to regular mango intake in OW/OB participants with chronic low grade inflammation. | Baseline to 4 weeks
  Fecal samples will be collected with standard collection kits and stored at -80°C until analysis. Metagenomic and transcriptomic analyses will be performed
Characterize indices of systemic inflammation (hs-CRP) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim will include analysis of systemic markers of inflammation (hs-CRP) in plasma
Characterize indices of systemic inflammation (TNF-α) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim will include analysis of systemic markers of inflammation (TNF-α) in plasma
Characterize indices of systemic inflammation (MCP-1) after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Assessments to address this aim will include analysis of systemic markers of inflammation (MCP-1) in plasma

SECONDARY OUTCOMES:
Characterize metabolite profiles after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Polyphenolic metabolites (phenolic acids and derivatives components) will be identified and quantified in urine and plasma.Metabolites in samples will be identified and quantified using an Agilent 6550 iFunnel UHPLC-QTOF-MS and6460 UHPLC-QQQ-MS, respectively
Assess insulin sensitivity after 4 week intake of mango beverage compared to a control beverage | Baseline to 4 weeks
  Insulin sensitivity assessment using oral glucose tolerance test (OGTT) method. Assessments to address this aim will include analysis of glucose and insulin concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Indika v, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No